CLINICAL TRIAL: NCT01726777
Title: Effect of Vitamin D Supplementation on Oral Glucose Tolerance in Subjects Exhibiting Marginal Vitamin D Status and an Increased Risk of Developing Diabetes.
Brief Title: Effect of Vitamin D Supplementation on Glucose Tolerance in Subjects at Risk for Diabetes With Low Vitamin D.
Acronym: EVIDENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dairy Farmers of Canada (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTRS-27546
Record Dates: First submitted 2012-11-09; First posted 2012-11-15 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes Mellitus; Vitamin D Deficiency
Keywords: Randomized controlled clinical trial; Diabetes; Vitamin D; Oral glucose tolerance; Blood glucose; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin D Deficiency; Diabetes Mellitus; Insulin Resistance | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): 30g normal cheddar cheese once per week
  Interventions: Dietary Supplement: Control
- Vitamin D (Experimental): 30g cheddar cheese containing 28,000IU vitamin D once per week
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Control — Normal cheddar cheese
  Arms: Control
Dietary Supplement: Vitamin D — Vitamin D3 supplemented cheddar cheese
  Other Names: Vitamin D3
  Arms: Vitamin D

SUMMARY:
Type 2 diabetes (T2D) is an increasingly common and serious condition. Studies show that low vitamin D levels are associated with increased diabetes risk and that vitamin D may protect against diabetes by reducing chronic inflammation and improving insulin sensitivity and insulin secretion. However, no studies have been able to show that vitamin D actually reduces post-prandial blood glucose levels, the most clinically relevant marker of diabetes. Previously the investigators have shown that cheddar cheese and low-fat cheese can be fortified with high levels of vitamin D and that this cheese is at least as a effective as vitamin D supplements in raising blood vitamin D levels.

The main purpose of this study is to see whether vitamin D enriched cheese can improve oral glucose tolerance (reduce blood glucose 2 hours after consuming a drink containing 75g sugar) in people who have low vitamin D levels and are at risk for developing T2D.

Other aims are to determine the effect of vitamin D may on insulin sensitivity, insulin secretion, markers of inflammation, blood cholesterol levels, and safety markers such as urinary calcium excretion.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is an increasingly prevalent and serious condition whose risk appears to be increased by low serum vitamin D concentrations. Epidemiological studies show an association between increased diabetes risk and low serum vitamin D and studies suggest that vitamin D may protect against diabetes by reducing chronic inflammation and improving insulin sensitivity and insulin secretion. Although clinical studies show some of these effects, no studies have been able to show that vitamin D supplementation reduces post-prandial blood glucose, the most clinically relevant marker of diabetes and dysglycemia. Previously, the investigators showed that cheddar cheese and low-fat cheese can be fortified with high levels of vitamin D3 (28,000IU/ 30g portion) and that, in this form, it is at least as a effective as vitamin D3 supplements in raising serum vitamin D concentrations. Since post-prandial glucose is most sensitive to changes in insulin sensitivity the main purpose of this study is to determine the effect of vitamin D supplementation on oral glucose tolerance (ie. serum glucose 2h after 75g oral glucose) in individuals who are at risk for developing T2D. Secondary objective are to determine the effect of vitamin D supplementation on insulin sensitivity, insulin secretion, inflammatory markers, blood lipids and markers of safety including serum parathyroid hormone levels and urinary calcium excretion.

ELIGIBILITY:
Inclusion Criteria:

* male or non-pregnant, non-lactating females, aged 18-75
* volunteered to participate by signing the consent form
* BMI <40kg/ m2
* vitamin D insufficient, defined as: serum 25(OH) vitamin D3 (25(OH)D) concentration ≤65nmol/ L
* increased risk for diabetes, defined as: FINDRISC score >10 for Caucasians or >6 for non-Caucasians OR presence of metabolic syndrome
* dysglycemia, defined as:fasting serum glucose 5.6 to 6.9 mmol/L, inclusive OR HbA1c 0.054 to 0.064, inclusive
* systolic blood pressure ≤150/95 mmHg if not being treated for hypertension or ≤140/90 mmHg if on treatment for hypertension.
* taking no prescription drugs, or stable (for at least 6 weeks) dose of birth control pill, or drug(s) used to treat hypertension, hyperlipidemia, depression or other mental illness or hypothyroid.
* taking no supplements, or stable (for at least 6 weeks) dose of supplement(s).

Exclusion Criteria:

* subjects not meeting all inclusion criteria
* history of renal failure or liver disease
* serum creatinine >1.8 times upper limit of normal (ULN)
* serum aspartate or alanine transaminase (AST,ALT) >3 times ULN
* current use of drug or drugs to treat diabetes or use of steroids or pancreatic enzymes
* within 6 weeks of randomization, change in dose of supplements or drug(s) used to treat hypertension, hyperlipidemia, depression or other mental illness or hypothyroid.
* use of antibiotics within 3 months.
* medical or surgical event requiring hospitalization within 3 months of randomization
* presence of any condition affecting nutrient absorption
* intolerance to cheese
* plan to travel outside Canada for more than 14 consecutive days during the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose concentration 2 hours after consuming 75g oral glucose (2 hour PC glucose, or 2hrPC glucose) | 24 Weeks
  Change from baseline in plasma glucose concentration 2 hours after consuming 75g oral glucose.

SECONDARY OUTCOMES:
Change in insulin resistance assessed using the homeostasis model assessment of insulin resistance (HOMA-IR) | 24 weeks
  Change from baseline in homeostasis model assessment of insulin resistance (HOMA-IR) which is G*I/22.5 where G is fasting plasma glucose (mmol/L) and I is fasting plasma insulin (uU/mL).
Change in Matsuda insulin sensitivity index | 24 weeks
  Change from baseline in Matsuda insulin sensitivity index which is (10,000/square root of [fasting glucose x fasting insulin] x [mean glucose x mean insulin during OGTT]).
Change in insulin secretion assessed using the homeostasis model assessment of beta-cell function (HOMA-B) | 24 weeks
  Change from baseline in homeostasis model assessment of beta-cell function (HOMA-B) which is 20*I/(G-3.5) where I is fasting plasma insulin (uU/mL) and G is fasting plasma glucose (mmol/L).
Change in insulinogenic index | 24 weeks
  Change from baseline in insulinogenic index which is dI0-30/dG0-30, where dI0-30 is the change in plasma insulin between fasting and 30min and dG0-30 is the change in plasma glucose between fasting and 30min after 75g oral glucose.
Change in disposition index derived from HOMA-IR and HOMA-B | 24 weeks
  Change from baseline in disposition index which is HOMA-B/HOMA-IR, which have been defined above.
Change in disposition index based on oral glucose tolerance test (OGTT) | 24 weeks
  Change from baseline in ISSI-2 index which is AUCi/AUCg x Matsuda insulin sensitivity index, where AUCi and AUCg, respectively, are the total areas under the plasma insulin and glucose response curves after 75g oral glucose and Matsuda insulin sensitivity index has been defined above.
Change in fasting plasma glucose | 24 weeks
  Change from baseline in fasting plasma glucose
Change in glucose area under the curve | 24 weeks
  Change from baseline in incremental area under the glucose response curve after 75g oral glucose
Change in glycated hemoglobin | 24 weeks
  Change from baseline in glycated hemoglobin (HbA1c)
Correlation between changes in serum 25-hydroxy-vitamin D concentration (25(OH)D) and changes in 2 hour PC glucose | 24 weeks
  Correlation between change from baseline in serum 25-hydroxy-vitamin D concentration and change from baseline in plasma glucose 2 hours after 75g oral glucose.

OTHER OUTCOMES:
Fasting serum 25(OH)D | 24 weeks
  Absolute concentration of serum 25-hydroxy-vitamin D3
Change in serum 25(OH)D | 24 weeks
  Change from baseline in serum 25-hydroxy-vitamin D3
Change in serum total cholesterol | 24 weeks
  Change from baseline in fasting serum total cholesterol
Change in serum low-density lipoprotein (LDL) cholesterol | 24 weeks
  Change from baseline in fasting serum calculated LDL cholesterol
Change in serum high-density lipoprotein (HDL) cholesterol | 24 weeks
  Change from baseline in fasting serum HDL cholesterol
Change in serum triglycerides | 24 weeks
  Change from baseline in fasting serum triglycerides
Change in serum apolipoprotein B (apoB) | 24 weeks
  Change from baseline in fasting serum apolipoprotein B
Change in serum c-reactive protein (CRP) | 24 weeks
  Change from baseline in fasting serum c-reactive protein
Change in serum orosomucoid | 24 weeks
  Change from baseline in fasting serum orosomucoid
Change in serum haptoglobin | 24 weeks
  Change from baseline in fasting serum haptoglobin
Change in serum alpha-1-antitrypsin | 24 weeks
  Change from baseline in fasting serum alpha-1-antitrypsin
Change in serum aspartate aminotransferase (AST) | 24 weeks
  Change from baseline in fasting serum aspartate aminotransferase
Change in serum alanine aminotransferase (ALT) | 24 weeks
  Change from baseline in fasting serum alanine aminotransferase
Serum calcium | 24 weeks
  Absolute concentration of serum calcium
Urinary calcium:creatinine ratio | 24 weeks
  Urinary calcium:creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, DM, PhD, Principal Investigator — University of Toronto
Locations (3):
- Canada (3):
  - University of Guelph, Guelph, Ontario
  - Glycemic Index Laboratories, Toronto, Ontario
  - Institut de recherches cliniques de Montréal, Montreal, Quebec